CLINICAL TRIAL: NCT05719025
Title: Markers of Neurological Damage Post Covid-19 in People Living With HIV (PLWH)
Brief Title: Markers of Neurological Damage Post Covid-19 in PLWH
Acronym: NeuroCOV-HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Paola Cinque, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: Neuro COV-HIV
Record Dates: First submitted 2022-10-18; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Hiv
MeSH Terms: conditions — COVID-19; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV + COVID+
- HIV + COVID -
- HIV - COVID +
- HIV- COVID-

SUMMARY:
Both HIV infection and Covid-19 are associated to cognitive and psychiatric impairment, like anxiety and depression. These disturbs are well-known in HIV infection and partially characterized in Covid-19.

DETAILED DESCRIPTION:
HIV has an high neurotropism and the HIV-associated dementia was one of the most frequent clinical complications and principal cause of death before the introduction of antiretroviral theraphy (ART). However, also in PLWH taking ART and with suppressed viral load over years, the proportion of neuro-cognitive impairment, anxiety and depression remain higher then the general population.

These problems may be the consequence of a persistent systemic and central nervous system (CNS) immuno-activation caused by the persistence of viral reservoir in the peripheric and tissutal lymphocytes.

Neurological and psychiatric problems have been described in a variable proportion in patients with corona virus disease 19 (COVID-19) and in the complex it doesn't seems to be the direct consequence of CNS cellular infection, but rather of inflammation and coagulations disorder due to COVID-19 in the nervous tissue.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ COVID+: people living with HIV that get corona virus disease 19 (COVID19) diagnosed at least 9 month ago with a positive rino-pharyngeal swab (molecular or antigenic), or with compatible clinic and a positive serologic test for Sars-CoV2 before the vaccination; Age > 50 years old, no gender.
* HIV+ COVID-: people living with HIV that had not get COVID19. Age>50 years; no gender.
* HIV- COVID+: people without HIV that get COVID19 diagnosed at least 9 month ago with a positive rino-pharyngeal swab (molecular or antigenic), or with compatible clinic and a positive serologic test for Sars-CoV2 before the vaccination; Age > 50 years old, no gender.
* HIV- COVID-: people without HIV that had not get COVID19 (healthy people and volunteers) Age>50 years; no gender.

Exclusion Criteria:

* Inability to perform the neuro-cognitive or functional tests due to neurologic deficit (inability to writing, reading, understand how to perform the tests)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * HIV+ COVID+: people living with HIV that get corona virus disease 19 (COVID19) diagnosed at least 9 month ago with a positive rino-pharingeal swab (molecular or antigenic), or with compatible clinic and a positive sierologic test for Sars-CoV2 before the vaccination; Age > 50 years old, no gender.
  * HIV+ COVID-: people living with HIV that had not get COVID19. Age>50 years; no gender.
  * HIV- COVID+: people without HIV that get COVID19 diagnosed at least 9 month ago with a positive rino-pharingeal swab (molecular or antigenic), or with compatible clinic and a positive sierologic test for Sars-CoV2 before the vaccination; Age > 50 years old, no gender.
  * HIV- COVID-: people without HIV that had not get COVID19 (healthy people and volunteers) Age>50 years; no gender.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Impact on neurological damage of COVID-19 in PLWH | Through study completion, an average of 1 year
  Assessing the impact of COVID-19 in PLWH concerning the neurological damage, by measuring blood's markers like the Neurofilament Light Protein (NfL) and the Glial Fibrillary Acidic Protein (gFAP)

SECONDARY OUTCOMES:
Frequency of neurocognitive and muscular (strength and balance) impairment | Through study completion, an average of 1 year
  Assessing the prevalence of: neurocognitive impairment, altered muscular function (strenght and balance), plasmatic level of Ubiquitin Carboxy-terminal Hydrolase L1 Neurons (UCH-L1) and total-tau, soluble and cellular infiammation's markers in blood and the expression profile of messenger ribonucleic acid (mRNA) in lymphocytes and the humoral and cellular answer against Sars-CoV2 in people living with HIV which had and ad not contract COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele Turro, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes